CLINICAL TRIAL: NCT06121492
Title: Oral Branched-chain Amino Acid Supplementation for Cirrhotic Patients With Sarcopenia: a Double-blinded Randomized Controlled Trial
Brief Title: Oral Branched-chain Amino Acid Supplementation for Cirrhotic Patients With Sarcopenia
Acronym: BCAASarcopenia
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI 655/2023
Record Dates: First submitted 2023-11-01; First posted 2023-11-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia; Cirrhosis of the Liver
Keywords: sarcopenia; cirrhosis; Branched-chain amino acids; nutrition
MeSH Terms: conditions — Sarcopenia; Fibrosis | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Intervention Model Description: The participants will be randomly and blindly divided into two groups: (branched-chain amino acids) BCAA group and the placebo group, using a 1:1 ratio, with each group consisting of 43 individuals. The blinded participants will take either BCAA or placebo for 24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All of participants, care providers, investigators and outcome assessors will be blinded. Only a research nurse will know which arm the participants are assigned to. The packages of BCAA and placebo are identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Branched-chain amino acid (Experimental): In the branched-chain amino acid (BCAA group), participants will receive oral BCAA for 24 weeks, with a daily dosage of approximately 13.68 g/day. Each sachet of BCAA will contain 6.84 g of BCAA (valine 1.82 g, leucine 3.29 g, isoleucine 1.72 g), total protein 17.08 g, carbohydrates 25.48 g, fat 5.66 g, providing 221.2 kcal of energy. Each sachet weighs 52 g and should be mixed with 150 ml of water. Participants will consume 2 sachets daily, one after breakfast and one after dinner.
  Interventions: Drug: Branched-chain amino acid
- Placebo (Placebo Comparator): In the placebo group, BCAA will be replaced with maltodextrin. Each sachet of the placebo will contain a total of 5.93 g of protein, 35.87 g of carbohydrates, 6.00 g of fat, providing 221.2 kcal of energy. Like the BCAA sachets, each placebo sachet will weigh 52 g and should be mixed with 150 ml of water. Participants in the placebo group will consume 2 sachets daily, one after breakfast and one after dinner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Branched-chain amino acid — In the BCAA group, participants will receive oral BCAA for 24 weeks, with a daily dosage of approximately 13.68 g/day. Each sachet of BCAA will contain 6.84 g of BCAA (valine 1.82 g, leucine 3.29 g, isoleucine 1.72 g), total protein 17.08 g, carbohydrates 25.48 g, fat 5.66 g, providing 221.2 kcal of energy. Each sachet weighs 52 g and should be mixed with 150 ml of water. Participants will consume 2 sachets daily, one after breakfast and one after dinner.
  Other Names: BCAA
  Arms: Branched-chain amino acid
Drug: Placebo — In the placebo group, BCAA will be replaced with maltodextrin. Each sachet of the placebo will contain a total of 5.93 g of protein, 35.87 g of carbohydrates, 6.00 g of fat, providing 221.2 kcal of energy. Like the BCAA sachets, each placebo sachet will weigh 52 g and should be mixed with 150 ml of water. Participants in the placebo group will consume 2 sachets daily, one after breakfast and one after dinner.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare the nutritional parameters after 24-week supplementation of branched-chain amino acids in cirrhotic patients with low muscle mass.

The main questions it aims to answer are:

Is there the differences in the proportions of cirrhotic patients recovering from low muscle mass at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there the differences in the change of skeletal muscle index (SMI) measured by abdominal computed tomography (CT) at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in other indices related to low muscle mass, including appendicular skeletal muscle mass (ASM), ASM/height^2, handgrip strength, and 6-meter walk speed at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in the liver frailty index (LFI), consisting of handgrip strength, chair stands, and balance, at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in serum albumin levels, at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in severity of liver disease, including the Model for End-Stage Liver Disease-Sodium Score (MELD-Na score), Child-Turcotte-Pugh score, and liver stiffness measured by transient elastography at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group?

Participants will be asked to do following tasks:

Participants will be asked for basic information such as age, place of residence, and contact phone number.

Participants will undergo measurements of body weight, height, body mass index (BMI), muscle mass, and body fat content using a body composition analyzer, a total of 2 times (at the beginning and end of the research), and an upper abdominal computed tomography (CT) scan without additional radiation exposure, only once (at the end of the research) throughout the study.

Participants will be tested for muscle function, including handgrip strength, a 6-meter walk test, chair stands, and balance, all performed twice (at the beginning and end of the research).

Laboratory testing will include a complete blood count, liver and kidney function, blood clotting function, mineral levels, cholesterol, and glucose. Blood will be drawn a total of 2 times (at the beginning and end of the research) during the study, with each blood draw approximately 15 milliliters (1 tablespoon).

Transient elastography will be performed twice (at the beginning and end of the research) during the study, with each Transient elastography taking approximately 10 minutes.

Participants will be randomly assigned to either the group receiving branched chain amino acid (BCAA) medication or the placebo group, and you will take the assigned medication twice daily for a total of 24 weeks.

Participants will receive dietary and exercise recommendations from the research team and nutritionists in a group format, taking approximately 1 hour.

Participants will have follow-up appointments to monitor your condition three times during the study, at weeks 4, 12, and 24. These appointments will include inquiries about side effects from medication and placebo use, exercise, and dietary intake, each lasting approximately 30 minutes.

Participants will be asked to take photos of your daily meals for 3 days before meeting with the physician at weeks 4 and 12, to provide data for assessing your calorie intake. Participants can send these meal images via the online application, prepared by our research team. If participants are unable to do so, participants will be asked to keep a food diary and report your food and portion sizes to the research team.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare the nutritional parameters after 24-week supplementation of branched-chain amino acids in cirrhotic patients with low muscle mass.

The main questions it aims to answer are:

Is there the differences in the proportions of cirrhotic patients recovering from low muscle mass at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there the differences in the change of skeletal muscle index (SMI) measured by abdominal computed tomography (CT) at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in other indices related to low muscle mass, including appendicular skeletal muscle mass (ASM), ASM/height^2, handgrip strength, and 6-meter walk speed at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in the liver frailty index (LFI), consisting of handgrip strength, chair stands, and balance, at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in serum albumin levels, at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group? Is there changes in severity of liver disease, including the Model for End-Stage Liver Disease-Sodium Score (MELD-Na score), Child-Turcotte-Pugh score, and liver stiffness measured by transient elastography at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group?

Participants will be asked to do following tasks:

Participants will be asked for basic information such as age, place of residence, and contact phone number.

Participants will undergo measurements of body weight, height, body mass index (BMI), muscle mass, and body fat content using a body composition analyzer, a total of 2 times (at the beginning and end of the research), and an upper abdominal computed tomography (CT) scan without additional radiation exposure, only once (at the end of the research) throughout the study.

Participants will be tested for muscle function, including handgrip strength, a 6-meter walk test, chair stands, and balance, all performed twice (at the beginning and end of the research).

Laboratory testing will include a complete blood count, liver and kidney function, blood clotting function, mineral levels, cholesterol, and glucose. Blood will be drawn a total of 2 times (at the beginning and end of the research) during the study, with each blood draw approximately 15 milliliters (1 tablespoon).

Transient elastography will be performed twice (at the beginning and end of the research) during the study, with each Transient elastography taking approximately 10 minutes.

Participants will be randomly assigned to either the group receiving branched chain amino acid (BCAA) medication or the placebo group, and you will take the assigned medication twice daily for a total of 24 weeks.

Participants will receive dietary and exercise recommendations from the research team and nutritionists in a group format, taking approximately 1 hour.

Participants will have follow-up appointments to monitor your condition three times during the study, at weeks 4, 12, and 24. These appointments will include inquiries about side effects from medication and placebo use, exercise, and dietary intake, each lasting approximately 30 minutes.

Participants will be asked to take photos of your daily meals for 3 days before meeting with the physician at weeks 4 and 12, to provide data for assessing your calorie intake. Participants can send these meal images via the online application, prepared by our research team. If participants are unable to do so, participants will be asked to keep a food diary and report your food and portion sizes to the research team.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85 years.
* Patients who have been diagnosed with liver cirrhosis due to any etiology.
* Patients with sarcopenia as determined by a computed tomography scan within the last 3 months. For males, sarcopenia is defined as a Skeletal Muscle Index (SMI) less than 42 cm²/m², and for females, an SMI less than 38 cm²/m²

Exclusion Criteria:

* Patients with hepatocellular carcinoma outside the Milan criteria.
* Patients with Overt Hepatic Encephalopathy or gastrointestinal bleeding within the last 6 months.
* Patients with refractory ascites (ascites that does not respond to treatment).
* Patients in the advanced stage of cirrhosis with Child-Turcotte-Pugh (CTP) score C.
* Patients with acute-on-chronic liver failure (ACLF).
* Patients with uncontrollable decompensated comorbidities, including chronic heart failure classified as NYHA 3-4, patients with kidney disease requiring dialysis, patients with severe obstructive lung disease classified as Gold D, patients with other non-liver cancers requiring chemotherapy, and patients with chronic infections such as tuberculosis.
* Patients who have previously undergone liver or kidney transplantation.
* Patients with Human Immunodeficiency Virus (HIV) infection.
* Pregnant or breastfeeding patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Resolution of sarcopenia | 24 weeks
  To study the differences in the proportions of patients with resolution from sarcopenia measured by abdominal computed tomography at 24 weeks among cirrhotic patients with sarcopenia who received BCAA supplementation and the placebo group for 24 weeks. Resolution of sarcopenia implies better nutritional status and prognosis.

SECONDARY OUTCOMES:
change of skeletal muscle index (SMI) measured by abdominal computed tomography (CT) | 24 weeks
  To study the differences in the change of skeletal muscle index (SMI, centimeter^2/meter^2) measured by abdominal computed tomography (CT) at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group
change of appendicular skeletal muscle mass (ASM) | 24 weeks
  To study changes in appendicular skeletal muscle mass (ASM, kg) measured by bioelectrical impedance at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Increase in appendicular skeletal muscle mass implies better nutritional status.
change of index of appendicular skeletal muscle mass (ASM, kg) divided by height squared (meter^2) | 24 weeks
  To study changes in index of appendicular skeletal muscle mass (ASM, kg) divided by height squared (meter^2) at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Increase index of appendicular skeletal muscle mass (ASM, kg) divided by height squared (meter^2) implies better nutritional status.
change of handgrip | 24 weeks
  To study changes in handgrip (kilograms) measured by digital handgrip strength dynamometer at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Increase in handgrip implies better physical performance.
change of 6-meter walk speed | 24 weeks
  To study changes in 6-meter walk speed (meter/second) at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Increase in 6-meter walk speed implies better nutritional status.
change of the liver frailty index (LFI) | 24 weeks
  To study changes in the liver frailty index (LFI), consisting of handgrip strength, chair stands, and balance, at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group.
change of serum albumin | 24 weeks
  To study changes in serum albumin levels (grams/deciliters), at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Increase in serum albumin implies better nutritional status.
change of MELD-Na score | 24 weeks
  To study changes in the Model for End-Stage Liver Disease-Sodium Score (MELD-Na score) at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Decrease of MELD-Na score implies improved severity of cirrhosis.
change of Child-Turcotte-Pugh score | 24 weeks
  To study changes in Child-Turcotte-Pugh score at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Decrease of Child-Turcotte-Pugh score implies improved severity of cirrhosis.
change of liver stiffness | 24 weeks
  To study changes in the liver stiffness (kPa) measured by transient elastography at 24 weeks among cirrhotic patients with low muscle mass who received BCAA supplementation and the placebo group. Decrease of liver stiffness implies improved severity of cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Phunchai Charatcharoenwitthaya, M.D., Principal Investigator — Mahidol University
Locations (1):
- Division of Gastroenterology, Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
To protect patients' confidentiality, we will not share individual participant data.

REFERENCES:
- [Background] Charatcharoenwitthaya P, Tansakul E, Chaiyasoot K, Bandidniyamanon W, Charatcharoenwitthaya N. Dietary Composition and Its Association with Newly Diagnosed Nonalcoholic Fatty Liver Disease and Insulin Resistance. Nutrients. 2021 Dec 11;13(12):4438. doi: 10.3390/nu13124438. PMID 34959990
- [Background] Sirisunhirun P, Bandidniyamanon W, Jrerattakon Y, Muangsomboon K, Pramyothin P, Nimanong S, Tanwandee T, Charatcharoenwitthaya P, Chainuvati S, Chotiyaputta W. Effect of a 12-week home-based exercise training program on aerobic capacity, muscle mass, liver and spleen stiffness, and quality of life in cirrhotic patients: a randomized controlled clinical trial. BMC Gastroenterol. 2022 Feb 14;22(1):66. doi: 10.1186/s12876-022-02147-7. PMID 35164698
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on nutrition in chronic liver disease. J Hepatol. 2019 Jan;70(1):172-193. doi: 10.1016/j.jhep.2018.06.024. Epub 2018 Aug 23. PMID 30144956
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Jaruvongvanich V, Thamtorawat S, Saiviroonporn P, Pisanuwongse A, Siriwanarangsun P. Sarcopenia as a Predictive Factor for Recurrence of Hepatocellular Carcinoma Following Radiofrequency Ablation. Asian Pac J Cancer Prev. 2023 Apr 1;24(4):1143-1150. doi: 10.31557/APJCP.2023.24.4.1143. PMID 37116135
- [Background] Mohta S, Anand A, Sharma S, Qamar S, Agarwal S, Gunjan D, Singh N, Madhusudhan KS, Pandey RM, Saraya A. Randomised clinical trial: effect of adding branched chain amino acids to exercise and standard-of-care on muscle mass in cirrhotic patients with sarcopenia. Hepatol Int. 2022 Jun;16(3):680-690. doi: 10.1007/s12072-022-10334-7. Epub 2022 Apr 25. PMID 35469091
- [Background] Siramolpiwat S, Limthanetkul N, Pornthisarn B, Vilaichone RK, Chonprasertsuk S, Bhanthumkomol P, Nunanan P, Issariyakulkarn N. Branched-chain amino acids supplementation improves liver frailty index in frail compensated cirrhotic patients: a randomized controlled trial. BMC Gastroenterol. 2023 May 15;23(1):154. doi: 10.1186/s12876-023-02789-1. PMID 37189033
- [Background] Hernandez-Conde M, Llop E, Gomez-Pimpollo L, Fernandez Carrillo C, Rodriguez L, Van Den Brule E, Perello C, Lopez-Gomez M, Abad J, Martinez-Porras JL, Fernandez-Puga N, Ferre C, Trapero M, Fraga E, Calleja JL. Adding Branched-Chain Amino Acids to an Enhanced Standard-of-Care Treatment Improves Muscle Mass of Cirrhotic Patients With Sarcopenia: A Placebo-Controlled Trial. Am J Gastroenterol. 2021 Nov 1;116(11):2241-2249. doi: 10.14309/ajg.0000000000001301. PMID 34074812
- [Background] Gluud LL, Dam G, Les I, Marchesini G, Borre M, Aagaard NK, Vilstrup H. Branched-chain amino acids for people with hepatic encephalopathy. Cochrane Database Syst Rev. 2017 May 18;5(5):CD001939. doi: 10.1002/14651858.CD001939.pub4. PMID 28518283
- [Background] Tajiri K, Shimizu Y. Branched-chain amino acids in liver diseases. Transl Gastroenterol Hepatol. 2018 Jul 30;3:47. doi: 10.21037/tgh.2018.07.06. eCollection 2018. PMID 30148232
- [Background] Soeters PB, Fischer JE. Insulin, glucagon, aminoacid imbalance, and hepatic encephalopathy. Lancet. 1976 Oct 23;2(7991):880-2. doi: 10.1016/s0140-6736(76)90541-9. PMID 62115
- [Background] Zenith L, Meena N, Ramadi A, Yavari M, Harvey A, Carbonneau M, Ma M, Abraldes JG, Paterson I, Haykowsky MJ, Tandon P. Eight weeks of exercise training increases aerobic capacity and muscle mass and reduces fatigue in patients with cirrhosis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1920-6.e2. doi: 10.1016/j.cgh.2014.04.016. Epub 2014 Apr 24. PMID 24768811
- [Background] Roman E, Torrades MT, Nadal MJ, Cardenas G, Nieto JC, Vidal S, Bascunana H, Juarez C, Guarner C, Cordoba J, Soriano G. Randomized pilot study: effects of an exercise programme and leucine supplementation in patients with cirrhosis. Dig Dis Sci. 2014 Aug;59(8):1966-75. doi: 10.1007/s10620-014-3086-6. Epub 2014 Mar 6. PMID 24599772
- [Background] Krell RW, Kaul DR, Martin AR, Englesbe MJ, Sonnenday CJ, Cai S, Malani PN. Association between sarcopenia and the risk of serious infection among adults undergoing liver transplantation. Liver Transpl. 2013 Dec;19(12):1396-402. doi: 10.1002/lt.23752. Epub 2013 Oct 21. PMID 24151041
- [Background] Tantai X, Liu Y, Yeo YH, Praktiknjo M, Mauro E, Hamaguchi Y, Engelmann C, Zhang P, Jeong JY, van Vugt JLA, Xiao H, Deng H, Gao X, Ye Q, Zhang J, Yang L, Cai Y, Liu Y, Liu N, Li Z, Han T, Kaido T, Sohn JH, Strassburg C, Berg T, Trebicka J, Hsu YC, IJzermans JNM, Wang J, Su GL, Ji F, Nguyen MH. Effect of sarcopenia on survival in patients with cirrhosis: A meta-analysis. J Hepatol. 2022 Mar;76(3):588-599. doi: 10.1016/j.jhep.2021.11.006. Epub 2021 Nov 14. PMID 34785325
- [Background] Li AA, Kim D, Ahmed A. Association of Sarcopenia and NAFLD: An Overview. Clin Liver Dis (Hoboken). 2020 Sep 4;16(2):73-76. doi: 10.1002/cld.900. eCollection 2020 Aug. No abstract available. PMID 32922754
- [Background] Therakomen V, Petchlorlian A, Lakananurak N. Prevalence and risk factors of primary sarcopenia in community-dwelling outpatient elderly: a cross-sectional study. Sci Rep. 2020 Nov 11;10(1):19551. doi: 10.1038/s41598-020-75250-y. PMID 33177536
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Luengpradidgun L, Chamroonkul N, Sripongpun P, Kaewdech A, Tanutit P, Ina N, Piratvisuth T. Utility of handgrip strength (HGS) and bioelectrical impedance analysis (BIA) in the diagnosis of sarcopenia in cirrhotic patients. BMC Gastroenterol. 2022 Mar 30;22(1):159. doi: 10.1186/s12876-022-02236-7. PMID 35354434
- [Background] Nishikawa H, Shiraki M, Hiramatsu A, Moriya K, Hino K, Nishiguchi S. Japan Society of Hepatology guidelines for sarcopenia in liver disease (1st edition): Recommendation from the working group for creation of sarcopenia assessment criteria. Hepatol Res. 2016 Sep;46(10):951-63. doi: 10.1111/hepr.12774. PMID 27481650
- [Background] Santilli V, Bernetti A, Mangone M, Paoloni M. Clinical definition of sarcopenia. Clin Cases Miner Bone Metab. 2014 Sep;11(3):177-80. PMID 25568649